CLINICAL TRIAL: NCT02756299
Title: Patient Education and PAP Compliance in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 89513307/1009/309
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea; Positive Airway Pressure; Patient Education
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Training Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device and Standard Care (Active Comparator): Positive Airway Pressure Device and Standard Support
  Interventions: Other: Standard Support
- Device and Educational Care (Active Comparator): Positive Airway Pressure Device and Educational Support
  Interventions: Other: Educational Support

INTERVENTIONS:
Other: Educational Support — General information about OSA and PAP treatment at baseline and additional polysomnography chart viewing from both diagnostic and titration nights
  Arms: Device and Educational Care
Other: Standard Support — General information about OSA and PAP treatment at baseline
  Arms: Device and Standard Care

SUMMARY:
Obstructive sleep apnea (OSA) is a common disorder with serious complications. Positive airway pressure (PAP) is the first line treatment of OSA, which eliminates obstructive events, reduces daytime sleepiness, and improves quality of life, especially in those with excessive daytime sleepiness. However, despite the benefits of the PAP treatment, overall acceptance and adherence rates are not fully promising. Less is known regarding the PAP adherence rates in Turkey. In the current study, the researchers primarily addressed if an intensified patient education strategy including the polysomnography (PSG) charts viewing followed by frequent follow-ups would improve the compliance rates at long-term in patients with OSA.

DETAILED DESCRIPTION:
OSA is a common disorder with serious complications. PAP is the first line treatment of OSA, but overall acceptance and adherence rates are not fully promising. In the current study, the researchers primarily addressed if an intensified patient education strategy including the PSG charts viewing followed by frequent follow-ups would improve the compliance rates at long-term in patients with OSA.

METHOD:

This single-center, randomized, controlled study was conducted at the Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital in Istanbul between June 2014 and April 2015. Eligible OSA patients were randomized to Standard Support (SS) group (general information about OSA and PAP treatment at baseline), or to Educational Support (ES) group (additional polysomnography chart viewing from both diagnostic and titration nights). All patients were scheduled to five PAP control visits between 2 weeks and 6 months after the PAP prescription. Primary outcome was the PAP compliance (4 h/night for 70% of all the nights) at the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients with newly diagnosed obstructive sleep apnea (apnea-hypopnea index ≥5 events/h), who were offered PAP treatment.
* Must be able to give informed consent

Exclusion Criteria:

* Disabled to come to follow-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Positive Airway Pressure usage (hours/night) | 6 months
  Satisfactory device usage defined as minimum 4 hours of night during at least 70% of period based on the objective measures from the device

CONTACTS AND LOCATIONS:
Overall Officials: Sema Sarac, MD, Study Chair — Istanbul Sureyyapasa Chest Diseases and Chest Surgery Hospital

IPD SHARING:
Plan to Share IPD: No